CLINICAL TRIAL: NCT04934709
Title: Immediate Effects of Photobiomodulation Therapy Combined With Static Magnetic Field on the Subsequent Performance: a Randomized Crossover Triple-blinded Placebo-controlled Trial
Brief Title: Photobiomodulation Therapy Combined With Static Magnetic Field on the Subsequent Performance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nove de Julho (Other)
Responsible Party: Principal Investigator, Ernesto Cesar Pinto Leal Junior, Full professor, University of Nove de Julho
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 665332
Record Dates: First submitted 2021-06-10; First posted 2021-06-22 (Actual); Last update posted 2021-06-22 (Actual); Status verified 2021-06

CONDITIONS: Skeletal Muscle Performance
Keywords: Photobiomodulation Therapy; Static Magnetic Field; Subsequent performance

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: A researcher programmed the device (placebo or PMBT-sMF) and was instructed not to inform the volunteers or other researchers as to the type of treatment (placebo or PBMT-sMF). Therefore, the researcher responsible for the treatment was blinded to the type of treatment administered to the volunteers. The sounds and signals emitted from the device as well as the information displayed on the screen was identical, regardless of the type of treatment (placebo or PBMT).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- PBMT-sMF (Experimental): Volunteers underwent intervention (active PBMT-sMF) in the non-dominant lower limb. A single application was performed at each phase of the trial, between the first and second set of the exercise protocol.
  Interventions: Device: Active PBMT-sMF
- Placebo (Placebo Comparator): Volunteers underwent intervention (placebo PBMT-sMF) in the non-dominant lower limb. A single application was performed at each phase of the trial, between the first and second set of the exercise protocol.
  Interventions: Device: Placebo PBMT-sMF

INTERVENTIONS:
Device: Active PBMT-sMF — PBMT-sMF was applied employing the Multi Radiance Medical Super Pulsed Laser MR4 console (Solon, Ohio, USA) with a LaserShower cluster probe as emitter. Six different sites of the knee extensor muscles (two medial, two lateral and two central points) were irradiated at the same time.
  Arms: PBMT-sMF
Device: Placebo PBMT-sMF — Placebo PBMT-sMF was applied employing the Multi Radiance Medical Super Pulsed Laser MR4 console (Solon, Ohio, USA) with a LaserShower cluster probe as emitter, but without any emission of therapeutic dose. Placebo PBMT-sMF was applied at six different sites of the knee extensor muscles (two medial, two lateral and two central points).
  Arms: Placebo

SUMMARY:
There is evidence about the effects of photobiomodulation therapy (PBMT) alone and combined with static magnetic field (PBMT-sMF) on skeletal muscle fatigue, physical performance and post-exercise recovery in different types of exercise protocols and sports activity. However, it is unknown the effects of PBMT-sMF to improve the subsequent performance after a first set of exercise. Therefore, the aim of this study was to investigate the effects of PBMT-sMF, applied between two sets of exercises, on the subsequent physical performance.

DETAILED DESCRIPTION:
A randomized, crossover, triple-blinded (assessors, therapist and volunteers), placebo-controlled trial was carried out. Healthy non-athletes' male volunteers were randomized and treated with a single application of PBMT-sMF and placebo between two sets of an exercise protocol performed on isokinetic dynamometer.

The order of interventions was randomized.

The primary outcome was fatigue index, measured by isokinetic dynamometer during the exercise protocol. The secondary outcomes were total work and peak torque measured by isokinetic dynamometer during the exercise protocol; and blood lactate, measured by blood samples collected before, 3 minutes after the first set of the exercise protocol, 3 minutes after the application of the intervention and 3 minutes after the second set of the exercise protocol.

Statistical analysis:

The findings were tested for normality using the Kolmogorov-Smirnov test and were determined to have a normal distribution. Data were expressed as the mean and standard deviation, and a two-way repeated measures ANOVA was performed to test between-group differences at each timepoint (treatment effects), mean difference (MD) and 95% confidence intervals (CI), followed by the Bonferroni post hoc test. The significance level was set at p < 0.05.

ELIGIBILITY:
Inclusion criteria:

* Male healthy volunteers;
* Non-athletes or those who practiced physical activity up to once a week;
* Aged 18-35 years.

Exclusion criteria

* History of musculoskeletal injuries in the hip and knee regions in the two months prior to the study;
* Use of pharmacological agents and nutritional supplements;
* Chronic joint disease in the non-dominant lower limb.

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2015-05 (Actual); Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Fatigue index | 1 minute after the end of exercise protocol.
  Variable provided directly by the isokinetic dynamometer during the exercise protocol.

SECONDARY OUTCOMES:
Total work | 1 minute after the end of exercise protocol.
  Variable provided directly by the isokinetic dynamometer during the exercise protocol.
Peak torque | 1 minute after the end of exercise protocol.
  Variable provided directly by the isokinetic dynamometer during the exercise protocol.
Blood lactate | 3 minutes after the first set of the exercise protocol, 3 minutes after the application of the intervention and 3 minutes after the second set of the exercise protocol.
  Measured by blood samples.

CONTACTS AND LOCATIONS:
Locations (1):
- Laboratory of Phototherapy and Innovative Technologies in Health, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Yes
Data will be shared upon request addressed to the principal investigator.
Supporting Information: Study Protocol, SAP, CSR